CLINICAL TRIAL: NCT04811716
Title: A Randomized, Open-label, Two-arm Study to Evaluate the Safety, Efficacy, and Pharmacodynamic Effects of Pozelimab and Cemdisiran Combination Treatment in Patients With Paroxysmal Nocturnal Hemoglobinuria Who Have Received Pozelimab Monotherapy
Brief Title: Pozelimab and Cemdisiran Combination Treatment in Adult Participants With Paroxysmal Nocturnal Hemoglobinuria Who Have Received Pozelimab Monotherapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R3918-PNH-2092; 2020-005005-17 (EudraCT Number)
Record Dates: First submitted 2021-03-19; First posted 2021-03-23 (Actual); Results first posted 2025-01-16 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: PNH
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Pozelimab Q4W + Cemdisiran (Experimental)
  Interventions: Drug: Pozelimab; Drug: Cemdisiran
- Pozelimab Q2W + Cemdisiran (Experimental)
  Interventions: Drug: Pozelimab; Drug: Cemdisiran

INTERVENTIONS:
Drug: Pozelimab — Administered Sub-cutaneous (SC) per protocol
  Other Names: REGN3918
Drug: Cemdisiran — Administered SC per protocol
  Other Names: ALN-CC5

SUMMARY:
The primary objective of the study is to evaluate the safety and tolerability of 2 dosing regimens of pozelimab and cemdisiran combination therapy during the open-label treatment period (OLTP)

The secondary objectives of the study are:

* To evaluate the effect of the combination treatment on the following parameters of intravascular hemolysis: lactate dehydrogenase (LDH) control, breakthrough hemolysis, and inhibition of total complement hemolysis activity (CH50)
* To evaluate the effect of the combination treatment on hemoglobin levels
* To evaluate the effect of the combination treatment on red blood cell (RBC) transfusion requirements
* To evaluate the effect of the combination treatment on clinical outcome assessments (COAs) measuring fatigue and health related quality of life
* To assess the concentrations of total pozelimab in serum and total complement component (C) 5 and cemdisiran in plasma
* To assess immunogenicity to pozelimab and cemdisiran
* To evaluate the long-term safety and efficacy of pozelimab and cemdisiran in an optional open-label extension period (OLEP)
* To assess safety after treatment intensification with pozelimab and cemdisiran

ELIGIBILITY:
Key Inclusion Criteria:

1. Participants with PNH who are receiving treatment with pozelimab monotherapy in the R3918- PNH-1868 study (NCT04162470)

Key Exclusion Criteria:

1. Documented, positive polymerase chain reaction (PCR) or equivalent test based on regional recommendations for COVID-19 or suspected SARS-CoV-2 infection as defined in the protocol
2. Participants with documented history of liver cirrhosis or participants with liver disease with evidence of currently impaired liver function; or participants with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) as described in the protocol
3. Significant protocol deviation(s) in the parent study based on the investigator's judgment as described in the protocol
4. Any new condition or worsening of an existing condition which, in the opinion of the investigator, would make the participant unsuitable for enrollment or would jeopardize the safety of the participant
5. Known hypersensitivity to cemdisiran or any component of cemdisiran formulation

NOTE: Other protocol-defined Inclusion/ Exclusion Criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2021-07-29 (Actual); Primary Completion 2022-10-25 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals
Locations (13):
- Prince of Wales Hospital, Hong Kong, New Territories, Hong Kong
- D l Pesti Centrumk rh z Orsz gos Hematol giai s Infektol giai Int zet, Budapest, Nagyvárad Tér 1, Hungary
- Malaysia (3):
  - Hospital Miri, Miri, Sarawak
  - Hospital Sibu, Sibu, Sarawak
  - Hospital Sultanah Nur Zahirah, Kuala Terengganu, Terengganu
- South Korea (5):
  - Samsung Medical Center, Seoul, Seoul Teugbyeolsi
  - Pusan National University Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Yonsei University College of Medicine, Severance Hospital, Seoul
  - Ewha Womans University Medical Centre, Seoul
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- St. James's University Hospital, Leeds, West Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/

REFERENCES:
- [Derived] Jang JH, Wong RSM, Hartford C, Pavani R, Aurand L, Nguyen Q, Mohan K, Meagher K, Sherman S, Rofail D, Perlee L, Souttou A, Kelly RJ. Safety, Efficacy, and Patient-Reported Outcomes From a Phase 2 Randomized Trial of Pozelimab and Cemdisiran Combination in Patients With Paroxysmal Nocturnal Hemoglobinuria. EJHaem. 2025 Jul 24;6(4):e70095. doi: 10.1002/jha2.70095. eCollection 2025 Aug. PMID 40708708
- See also: A Plain Language Summary is available on TrialSummaries.com — https://www.trialsummaries.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Twenty-four participants were screened and randomized.
Groups:
- Pozelimab Q2W + Cemdisiran: Pozelimab administered by subcutaneous (SC) injection every 2 weeks (Q2W) and cemdisiran administered by subcutanous (SC) injection. The first dose of the combination treatment (pozelimab Q2W + cemdisiran) was administered on day 1 of the open-label treatment period (OLTP). In the open- label extension period (OLEP), participants received a regimen of pozelimab + cemdisiran, regardless of their treatment assignment in the OLTP.
- Pozelimab Q4W + Cemdisiran: Pozelimab administered by subcutaneous (SC) injection every 4 weeks (Q4W) and cemdisiran administered by subcutanous (SC) injection. The first dose of the combination treatment was administered on day 1 of the OLTP. In the OLEP, participants received a regimen of pozelimab Q4W + cemdisiran, regardless of their treatment assignment in the OLTP.
Period: Overall Study
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Started | 12 | 12
Completed | 10 | 12
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.4 (16.89) | 53.2 (16.38) | 47.3 (17.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 11
  Male | 7 | 6 | 13
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  Asian | 10 | 11 | 21
  American Indian or Alaska Native | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Open Label Treatment Period (OLTP)
Time Frame: Through Week 28
Population: Safety analysis set (SAF) included all randomized participants who received any amount of study drug and was based on the treatment received (as treated); Here 'number analyzed' = the number of evaluable participants at a specified timepoint
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants
  Participants with any TEAE | 66.7 | 41.7
  Participants with serious TEAE | 16.7 | 0
  Participants with severe TEAE | 16.7 | 0

2. Secondary Outcome: Percent Change of Lactate Dehydrogenase (LDH) From Pre-treatment to End-of-treatment Period
Description: OLTP Pre-treatment (mean of LDH values prior to combination dosing); End-of-treatment (mean of LDH value at week 24- through week 28); percentage of change in Upper Limit of Normal (xULN).
Time Frame: End of treatment period, approximately 28 Weeks
Population: Full analysis set (FAS) = included all randomized participants who received any amount of study drug & had at least 1 post-baseline assessment; based on treatment allocated (as randomized); Here 'number analyzed' = number of evaluable participants at a specified timepoint
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of change | 2.93 (36.575) | 3.65 (13.608)

3. Secondary Outcome: Percentage of Participants Maintaining Adequate Control of Hemolysis From Baseline (Day 1) Through Week 28
Description: OLTP Adequate control of hemolysis is defined as LDH values ≤1.5 × Upper limit of normal (ULN) from baseline (day 1) to week 28
Time Frame: Baseline (Day 1) through Week 28
Population: Full analysis set (FAS) = included all randomized participants who received any amount of study drug & had at least 1 post-baseline assessment; based on treatment allocated (as randomized); Here 'number analyzed' is the number of evaluable participants at a specified timepoint
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants | 75.0 | 91.7

4. Secondary Outcome: Percentage of Participants Maintaining Adequate Control of Hemolysis From Week 4 Through Week 28
Description: OLTP
Time Frame: Week 4 through Week 28
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of Participants | 83.3 | 91.7

5. Secondary Outcome: Percentage of Participants With Adequate Control of Hemolysis at Each Visit Day 1 Through Week 28
Description: OLTP; Adequate control at a visit is defined as having LDH <=1.5 x ULN at that visit
Time Frame: Day 1 through Week 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants
  Baseline Visit (Day 1) | 100.0 | 100.0
  Pre-treatment | 100.0 | 100.0
  Week 1 | 100.0 | 100.0
  Week 2 | 100.0 | 100.0
  Week 4 | 83.0 | 100.0
  Week 6 | 92.0 | 100.0
  Week 8: number analyzed (Participants) | 12 | 11
  Week 8 | 100.0 | 100.0
  Week 10: number analyzed (Participants) | 11 | 12
  Week 10 | 100.0 | 100.0
  Week 12 | 100.0 | 92.0
  Week 16 | 100.0 | 100.0
  Week 20 | 100.0 | 100.0
  Week 24 | 100.0 | 100.0
  Week 28 | 92.0 | 100.0

6. Secondary Outcome: Percentage of Participants With Normalization of LDH at Each Visit From Baseline (Day 1) Through Week 28
Description: OLTP; Normalization of LDH was defined as LDH ≤1.0 × ULN at each visit
Time Frame: Baseline (Day 1) through Week 28
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants
  Baseline (Day 1) | 92.0 | 75.0
  Pre-treatment | 92.0 | 83.0
  Week 1 | 100.0 | 92.0
  Week 2 | 92.0 | 83.0
  Week 4 | 83.0 | 83.0
  Week 6 | 83.0 | 75.0
  Week 8: number analyzed (Participants) | 12 | 11
  Week 8 | 100.0 | 82.0
  Week 10: number analyzed (Participants) | 11 | 12
  Week 10 | 100.0 | 83.0
  Week 12 | 92.0 | 83.0
  Week 16 | 92.0 | 75.0
  Week 20 | 100.0 | 92.0
  Week 24 | 100.0 | 92.0
  Week 28 | 83.0 | 83.0

7. Secondary Outcome: Average LDH (U/L) Based on Area Under the Curve (AUC) From OLTP Baseline (Day 1) Through Week 28
Description: OLTP
Time Frame: Baseline (Day 1) through Week 28
Population: Full analysis set (FAS) = included all randomized participants who received any amount of study drug & had at least 1 post-baseline assessment; based on treatment allocated (as randomized); Here 'n' = the number of evaluable participants at a specified timepoint
Measure: Mean (Standard Deviation); unit: Units per Liter (U/L)
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Units per Liter (U/L) | 238.18 (44.006) | 244.42 (39.085)

8. Secondary Outcome: Average LDH (U/L) Based on Area Under the Curve (AUC) From OLTP Week 4 Through Week 28
Description: OLTP
Time Frame: Week 4 through Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
U/L | 202.49 (38.272) | 211.28 (34.280)

9. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis From Baseline (Day 1) Through Week 28
Description: OLTP
  Breakthrough hemolysis is defined as an increase in LDH with concomitant signs or symptoms associated with hemolysis:
  • An increase in LDH occurs when:
  * LDH ≥2 × ULN if pre-treatment LDH is ≤1.5 × ULN or
  * LDH ≥2 × ULN after initial achievement of LDH ≤1.5 × ULN if pre-treatment LDH is >1.5 × ULN Signs or symptoms should correspond to those known to be associated with intravascular hemolysis due to Paroxysmal nocturnal hemoglobinuria (PNH) limited to the following: new onset or worsening fatigue, headache, dyspnea, hemoglobinuria, abdominal pain, scleral icterus, erectile dysfunction, chest pain, confusion, dysphagia, anemia including hemoglobin value significantly lower (ie, ≥2g/dL decrease) compared to patient's known baseline hemoglobin values, and thrombotic event.
Time Frame: Baseline (Day 1) through Week 28
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants | 8.3 | 0.0

10. Secondary Outcome: Percentage of Participants With Hemoglobin Stabilization From Baseline (Day 1) Through Week 28
Description: OLTP Hemoglobin stabilization was defined as participants who did not receive an RBC transfusion and had no decrease in hemoglobin level of ≥2 grams per deciLiter (g/dL).
Time Frame: Baseline (Day 1) through Week 28
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants | 75.0 | 91.7

11. Secondary Outcome: Change in Hemoglobin Levels From Baseline (Day 1) Through Week 28
Description: OLTP
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: grams per Liter (g/L)
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 11 | 12
grams per Liter (g/L) | -1.3 (13.77) | 10.3 (7.41)

12. Secondary Outcome: Percentage of Participants With Transfusion Avoidance From Baseline (Day 1) Through Week 28
Description: OLTP Not requiring a red blood cell (RBC) transfusion as per protocol algorithm
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Percentage of participants | 83.3 | 100.0

13. Secondary Outcome: Rate of Red Blood Cells (RBCs) Transfused From Baseline (Day 1) to Week 28
Description: OLTP Rate of RBCs transfused is defined as number of events per person-years of treatment. For each participant, the participant-years are the time from first dose date to week 28 (or early terminations visit if subject discontinued the study early) in the OLTP.
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Events per person-years of treatment
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Events per person-years of treatment | 1.284 [0.169 to 9.760] | NA [NA to NA] — No per-protocol transfusions occurred in the Q4W arm

14. Secondary Outcome: Number of Per-Protocol RBC Units Transfused From Baseline (Day 1) Through Week 28
Description: OLTP
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Units | 1.5 (3.73) | 0.0 (0.00)

15. Secondary Outcome: Change in Total Complement Hemolysis Activity Assay (CH50) From Baseline (Day 1) Through Week 28
Description: OLTP
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Units per milliliter (U/mL)
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Units per milliliter (U/mL) | 0.0 (0.0) | -0.1 (0.29)

16. Secondary Outcome: Change in Fatigue as Measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale From Baseline (Day 1) Through Week 28
Description: OLTP FACIT fatigue is a 13-item scale and for each item 4 is not at all fatigued to 0 very much fatigued. Higher FACIT-Fatigue scores indicate less fatigue (scores range from 0-52). A 5-point change is considered clinically meaningful.
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 8 | 9
Score on a scale | -6.0 (10.09) | -2.0 (4.36)

17. Secondary Outcome: Change in Global Health Status/Quality of Life Scale (GHS/QoL) on the European Organization for Research and Treatment of Cancer: Quality-of-Life Questionnaire Core 30 Items (EORTC QLQ-C30) From Baseline (Day 1) Through Week 28
Description: OLTP EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. Items contributing to the GHS/QoL, were scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that transformed score lies between 0 to 100. A higher score indicates better global health status/functioning and a negative change from baseline indicated less improvement.
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 8 | 9
Score on a scale | -9.4 (23.33) | -1.9 (13.03)

18. Secondary Outcome: Change in Physical Function (PF) Scores on the EORTC QLQ-C30 From Baseline (Day 1) Through Week 28
Description: OLTP; EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. Items contributing to the GHS/QoL, were scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that transformed score lies between 0 to 100. A higher score indicates better global health status/functioning and a negative change from baseline indicated less improvement.
Time Frame: Baseline (Day 1) to Week 28
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 8 | 9
Score on a scale | -6.7 (19.19) | 0.7 (9.09)

19. Secondary Outcome: Concentrations of Total Pozelimab in Serum on Week 28
Description: OLTP
Time Frame: On Week 28
Population: The pharmacokinetic (PK) analysis set includes all treated participants who received any amount of study drug (SAF) and who had at least 1 non-missing analyte measurement following the first dose of combination treatment. The PK analysis set is based on the actual treatment received.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
mg/L | 131 (74.8) | 58.2 (31.5)

20. Secondary Outcome: Concentrations of Cemdisiran in Plasma on Week 28
Description: OLTP
Time Frame: On Week 28
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
mg/L | NA (NA) — There were no quantifiable concentration at this time point | NA (NA) — There were no quantifiable concentration at this time point

21. Secondary Outcome: Concentrations of Total C5 on Week 28
Description: OLTP
Time Frame: On Week 28
Population: as for outcome 19
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
mg/L | 0 [0 to 13.8] | 0 [0 to 0]

22. Secondary Outcome: Number of Participants With Pozelimab Anti-Drug Antibody (ADA) Responses Over Time
Description: OLTP and OLEP
Time Frame: Up to Week 52 (OLTP [ Week 0 - Week 28] + OLEP [Week 28 - Week 52])
Population: Anti-Drug Antibodies (ADA) Analysis Set; Here 'n' = the number of evaluable participants at a certain timepoint
Measure: Number; unit: Participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Participants
  Treatment-Boosted Response | 0 | 0
  Treatment-Emergent Response | 0 | 0

23. Secondary Outcome: Number of Participants With Cemdisiran Anti-Drug Antibody (ADA) Responses Over Time
Description: OLTP and OLEP
Time Frame: Up to Week 52 (OLTP [ Week 0 - Week 28] + OLEP [Week 28 - Week 52])
Population: Anti-Drug Antibodies (ADA) Analysis Set; Here 'n' = the number of evaluable participants at a certain timepoint
Measure: Number; unit: Participants
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
Participants
  Treatment-Boosted Response | 0 | 0
  Treatment-Emergent Response | 0 | 1

24. Secondary Outcome: Percentage of Participants With TEAEs for Participants Who Received Treatment Intensification
Description: OLTP No participants received dose intensification during the study; Therefore, assessment of the safety of pozelimab + cemdisiran combination therapy in participants requiring dose intensification was not conducted.
Time Frame: Through Week 28
Population: Safety analysis set (SAF) included all randomized participants who received any amount of study drug and was based on the treatment received (as treated); Here 'n' = the number of evaluable participants at a specified timepoint
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 0 | 0

25. Secondary Outcome: Change of LDH From Baseline (Day 1e) to Week 24e
Description: Optional Open-Label Extension Period (OLEP)
Time Frame: Baseline (Day 1e) to Week 24e
Population: OLEP FAS included all participants who participated in the OLEP who received any amount of study drug in the OLEP and had at least 1 post-baseline efficacy assessment in the OLEP; Here 'n' = number of evaluable participants at a specified timepoint
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 22
U/L | -18.2 (108.40)

26. Secondary Outcome: Percent Change of LDH From OLEP Baseline (Day 1e) to Week 24e
Description: OLEP; Percentage of change for units per liter (U/L)
Time Frame: Baseline (Day 1e) to Week 24e
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 22
Percentage of change | -0.7 (20.60)

27. Secondary Outcome: Change of LDH From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 22
U/L | -14.5 (105.90)

28. Secondary Outcome: Percent Change of LDH From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 22
Percentage of change | 0.2 (19.49)

29. Secondary Outcome: Percentage of Participants Maintaining Adequate Control of Hemolysis From Baseline (Day 1e) Through Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) through Week 24e
Population: OLEP FAS included all participants who participated in the OLEP who received any amount of study drug in the OLEP and had at least 1 post-baseline efficacy assessment in the OLEP; Here 'n' = the number of evaluable participants at a specified timepoint
Measure: Number; unit: Percentage of Participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of Participants | 95.7

30. Secondary Outcome: Percentage of Participants Maintaining Adequate Control of Hemolysis From Baseline (Day 1e) Through Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) through Week 52e
Population: as for outcome 25
Measure: Number; unit: Percentage of Participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of Participants | 95.7

31. Secondary Outcome: Percentage of Participants With Adequate Control of Hemolysis at Each Visit From Baseline (Day 1e) Through Week 52e
Description: OLEP Adequate control at a visit is defined as having LDH <=1.5 x ULN at that visit
Time Frame: Baseline (Day 1e) through Week 52e
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of participants
  OLEP Baseline (Day 1e) | 96.0
  Week 8e | 100.0
  Week 16e | 100.0
  Week 24e | 100.0
  Week 32e | 100.0
  Week 40e | 100.0
  Week 52e | 100.0

32. Secondary Outcome: Percentage of Participants With Normalization of LDH at Each Visit From Baseline (Day 1e) Through Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) through week 52e
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of participants
  OLEP Baseline (Day 1e) | 87.0
  Week 8e | 83.0
  Week 16e | 82.0
  Week 24e | 82.0
  Week 32e | 86.0
  Week 40e | 82.0
  Week 52e | 82.0

33. Secondary Outcome: Average LDH (U/L) Based on Area Under the Curve (AUC) From OLEP Baseline (Day 1e) Through Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) through Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
U/L | 154.63 (38.231)

34. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis From Baseline (Day 1e) Through Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) through Week 24e
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of Participants | 4.3

35. Secondary Outcome: Percentage of Participants With Breakthrough Hemolysis From Baseline (Day 1e) Through Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) through Week 52e
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of participants | 4.3

36. Secondary Outcome: Percentage of Participants With Hemoglobin Stabilization From Baseline (Day 1e) Through Week 24e
Description: OLEP Participants who did not receive RBC transfusion and had no decrease in hemoglobin levels
Time Frame: Baseline (Day 1e) through Week 24e
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of participants | 78.3

37. Secondary Outcome: Percentage of Participants With Hemoglobin Stabilization From Baseline (Day 1e) Through Week 52e
Description: OLEP Participants who did not receive RBC transfusion and had no decrease in hemoglobin levels
Time Frame: Baseline (Day 1e) through Week 52e
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of participants | 69.6

38. Secondary Outcome: Change in Hemoglobin Levels From Baseline (Day 1e) to Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 24e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 21
g/L | 0.8 (15.63)

39. Secondary Outcome: Change in Hemoglobin Levels From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 22
g/L | -0.6 (12.60)

40. Secondary Outcome: Percentage of Participants With Per-Protocol Transfusion Avoidance From Baseline (Day 1e) Through Week 24e
Description: OLEP Not requiring a RBC transfusion as per protocol algorithm
Time Frame: Baseline (Day 1e) through Week 24e
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of Participants | 87.0

41. Secondary Outcome: Percentage of Participants With Per-Protocol Transfusion Avoidance From Baseline (Day 1e) Through Week 52e
Description: OLEP Not requiring a RBC transfusion as per protocol algorithm
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Number; unit: Percentage of Participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of Participants | 87.0

42. Secondary Outcome: Rate of RBCs Transfused From Baseline (Day 1e) to Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 24e
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: Events per person-years of treatment
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Events per person-years of treatment | 0.591 [0.143 to 2.445]

43. Secondary Outcome: Rate of RBCs Transfused From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Number (95% Confidence Interval); unit: Events per person-years of treatment
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Events per person-years of treatment | 0.506 [0.092 to 2.773]

44. Secondary Outcome: Number of Units of RBCs Transfused From Baseline (Day 1e) to Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 24e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Units | 0.4 (1.47)

45. Secondary Outcome: Number of Units of RBCs Transfused From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Units
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Units | 0.9 (3.95)

46. Secondary Outcome: Change in CH50 From Baseline (Day 1e) to Week 16e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 16e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
U/mL | 0.0 (0.00)

47. Secondary Outcome: Change in CH50 From Baseline (Day 1e) to Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 24e
Population: OLEP FAS included all participants who participated in the OLEP who received any amount of study drug in the OLEP and had at least 1 post-baseline efficacy assessment in the OLEP; Here 'n' = the number of evaluable participants at a specified timepoint; No CH50 samples were collected at Week 24e
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 0

48. Secondary Outcome: Change in CH50 From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: U/mL
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 22
U/mL | 0.0 (0.21)

49. Secondary Outcome: Percent Change in CH50 From Baseline (Day 1e) to Week 16e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 16e
Population: OLEP FAS included all participants who participated in the OLEP who received any amount of study drug in the OLEP and had at least 1 post-baseline efficacy assessment in the OLEP; Here 'n' = the number of evaluable participants at a specified timepoint; Since all participants had 0 values at baseline for CH50, the percentage change was not appropriate and undefined. Therefore, this endpoint was not able to be calculated.
Measure: Number; unit: Percentage of change
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of change | NA — All participants had values of 0 at baseline for CH50, the percentage change was not appropriate and undefined

50. Secondary Outcome: Percent Change in CH50 From Baseline (Day 1e) to Week 24e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 24e
Population: OLEP FAS included all participants who participated in the OLEP who received any amount of study drug in the OLEP and had at least 1 post-baseline efficacy assessment in the OLEP; Here 'n' = number of evaluable participants at a specified timepoint; Since all participants had 0 values at baseline for CH50, the percentage change was not appropriate and undefined. Therefore, this endpoint was not able to be calculated.
Measure: Number; unit: Percentage of change
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of change | NA — All participants had values of 0 at baseline for CH50, the percentage change was not appropriate and undefined

51. Secondary Outcome: Percent Change in CH50 From Baseline (Day 1e) to Week 52e
Description: OLEP
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 49
Measure: Number; unit: Percentage of change
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of change | NA — All participants had values of 0 at baseline for CH50, the percentage change was not appropriate and undefined

52. Secondary Outcome: Change in Fatigue as Measured by Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-Fatigue) Scale From Baseline (Day 1e) to Week 52e
Description: OLEP; The FACIT-Fatigue is a 13-item, self-administered assessment of an individual's level of fatigue during their usual daily activities over the past week. This questionnaire is part of the FACIT measurement system, a compilation of questions measuring health-related QoL in participants with cancer and other chronic illnesses. The FACIT-Fatigue items are measured with a 5-point Likert scale ranging from 0 (not at all) to 4 (very much). Scores range from 0 to 52, with higher scores indicating less fatigue. A 5-point change is considered clinically meaningful.
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 21
Score on a scale | -0.9 (5.95)

53. Secondary Outcome: Change in GHS/QoL on the EORTC QLQ-C30 From Baseline (Day 1e) to Week 52e
Description: OLEP; EORTC QLQ-C30 is a 30-question tool used to assess the overall quality of life (QoL) in cancer participants. Items contributing to the GHS/QoL, were scored 1 ("very poor") to 7 ("excellent"). A linear transformation was applied to the raw scores so that transformed score lies between 0 to 100. A higher score indicates better global health status/functioning and a negative change from baseline indicated less improvement.
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 21
Score on a scale | 6.0 (13.73)

54. Secondary Outcome: Change in PF Scores on the EORTC QLQ-C30 From Baseline (Day 1e) to Week 52e
Description: as for outcome 53
Time Frame: Baseline (Day 1e) to Week 52e
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 21
Score on a scale | -0.3 (3.93)

55. Secondary Outcome: Percentage of Participants With TEAEs Up to Week 52
Description: OLEP
Time Frame: Up to Week 52
Population: The OLEP SAF includes all participants who participated in the OLEP who received any amount of study drug in the OLEP; Here 'n' = number of evaluable participants at a specified timepoint
Measure: Number; unit: Percentage of participants
Arm/Group | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 23
Percentage of participants
  Participants with any TEAE | 73.9
  Participants with serious TEAE | 8.7
  Participants with severe TEAE | 4.3

56. Secondary Outcome: Concentrations of Total Pozelimab in Serum on Week 52
Description: OLEP
Time Frame: On Week 52
Population: The OLEP pharmacokinetic (PK) analysis set includes all participants who participated in the OLEP who received any amount of study drug in the OLEP and who had at least 1 non-missing analyte measurement following the first dose of study drug in the OLEP.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
mg/L | 63.4 (35.6) | 58.6 (28.7)

57. Secondary Outcome: Concentrations of Total C5 on Week 52
Description: OLEP
Time Frame: On Week 52
Population: as for outcome 56
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
mg/L | 0 [0 to 8.05] | NA [NA to NA] — There were no quantifiable concentration at this time point

58. Secondary Outcome: Concentrations of Cemdisiran in Plasma on Week 52
Description: OLEP
Time Frame: On Week 52
Population: as for outcome 56
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Pozelimab Q2W + Cemdisiran | Pozelimab Q4W + Cemdisiran
Number analyzed (Participants) | 12 | 12
mg/L | NA (NA) — There were no quantifiable concentration at this time point | NA (NA) — There were no quantifiable concentration at this time point

ADVERSE EVENTS:
Time Frame: From first dose up to Week 52
Groups:
- OLTP_Pozelimab Q2W + Cemdisiran: Pozelimab administered by subcutaneous (SC) injection every 2 weeks (Q2W) and cemdisiran administered by subcutanous (SC) injection. The first dose of the combination treatment (pozelimab Q2W + cemdisiran) was administered on day 1 of the open-label treatment period (OLTP). In the open- label extension period (OLEP), participants received a regimen of pozelimab + cemdisiran, regardless of their treatment assignment in the OLTP.
- OLTP_Pozelimab Q4W + Cemdisiran: Pozelimab administered by subcutaneous (SC) injection every 4 weeks (Q4W) and cemdisiran administered by subcutanous (SC) injection. The first dose of the combination treatment was administered on day 1 of the OLTP. In the OLEP, participants received a regimen of pozelimab Q4W + cemdisiran, regardless of their treatment assignment in the OLTP.
- OLEP_Pozelimab Q4W + Cemdisiran: In the open-label extension period (OLEP), participants received a regimen of pozelimab SC Q4W + cemdisiran SC, regardless of their treatment assignment in the OLTP.
Arm/Group | OLTP_Pozelimab Q2W + Cemdisiran | OLTP_Pozelimab Q4W + Cemdisiran | OLEP_Pozelimab Q4W + Cemdisiran
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/23
Serious Adverse Events (participants affected / at risk) | 3/12 | 0/12 | 2/23
Other Adverse Events (participants affected / at risk) | 8/12 | 5/12 | 10/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLTP_Pozelimab Q2W + Cemdisiran (N=12) | OLTP_Pozelimab Q4W + Cemdisiran (N=12) | OLEP_Pozelimab Q4W + Cemdisiran (N=23)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OLTP_Pozelimab Q2W + Cemdisiran (N=12) | OLTP_Pozelimab Q4W + Cemdisiran (N=12) | OLEP_Pozelimab Q4W + Cemdisiran (N=23)
Injection site reaction (General disorders) | 2 (6) | 2 (4) | 3 (4)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 1 (1) | 4 (4)
Chlamydial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 4 (5)
Free haemoglobin present (Investigations) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram ST segment depression (Investigations) | 1 (1) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (2) | 0 (0) | 0 (0)
Breakthrough haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Inner ear disorder (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Paroxysmal nocturnal haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator has the right to independently publish study results from the investigator's site after a multi-center publication, or a defined period after the completion of the study by all sites. The investigator must provide the sponsor a copy of any such publication derived from the study for review and comment in advance of any submission, and delay publication, if requested, to allow the Sponsor to preserve its proprietary rights.

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04811716/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT04811716/SAP_001.pdf